CLINICAL TRIAL: NCT06365281
Title: Caries Prevalence, Experience and Risk Related Factors Among Early Middle-aged Patients Attending Faculty of Dentistry, Cairo University
Brief Title: Caries Prevalence, Experience and Risk Related Factors Among Early Middle-aged Patients Attending Cairo University
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohga Salah Fikry, principle investigator, Cairo University
Other Study IDs: CARIES PREVALENCE
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries; Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dental caries, a widespread oral health issue, results from a complex interplay of factors including behavior, hygiene, diet, and socio-demographic aspects. While preventive measures are available, it remains prevalent globally, affecting numerous teeth per individual. Improved oral hygiene practices and increased awareness have led to a reduction in caries prevalence. However, rising sugar consumption exceeds dietary guidelines, contributing to the problem. Despite limited epidemiological studies in Egypt, addressing individual-level factors is crucial. Surveillance of oral health in the early middle age group is standard, allowing decision-makers to assess the impact of caries and oral health care provision. Stratifying data by age, geography, and gender aids in understanding prevalence and planning effective prevention strategies. Overall, promoting awareness of dietary habits and preventive practices is vital for improving oral health outcome So, The purpose of this study is to assess the prevalence of dental caries among early middle age patients attending dental hospital in Faculty of Dentistry, Cairo university and to analyze the related risk factors utilizing WHO Oral Health Questionnaire for Adults.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age between 35 to 44 years old.
2. Patient consulting in the outpatient clinic
3. Provide informed consent
4. Co-operative patients approving to participate in the trial.
5. Males & Females
6. Egyptian

Exclusion Criteria:

1. Patients under or over this age group
2. Lack of compliance
3. Disabilities

Ages: 35 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Patients whose age between 35 to 44 years old.
  2. Patient consulting in the outpatient clinic
  3. Provide informed consent
  4. Co-operative patients approving to participate in the trial.
  5. Males & Females
  6. Egyptian
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental caries | 1 year
  DMFT index developed by World Health Organization (WHO) using numbered scores and percentge

SECONDARY OUTCOMES:
Caries experience | 1 year
  WHO severity criteria for adults 35-44 years of age , Very low <5.0 Low 5.0-8.9 Moderate 9.0-13.9 High >13.9
Caries risk related factors | 1 year
  WHO oral health questionnaire for adults 2013 (Dentist administrated)

CONTACTS AND LOCATIONS:
Overall Officials: Cairo University, Study Chair — Cairo University
Locations (1):
- Cairo university, Giza, Egypt